CLINICAL TRIAL: NCT03507920
Title: The Effects of Spinal Mobilizations on Neck Pain and Sympathetic Nervous System Activity in People With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10/2016/095
Record Dates: First submitted 2018-04-09; First posted 2018-04-25 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck passive mobilizations (Experimental)
  Interventions: Other: Neck passive mobilizations
- Manual contact (Placebo Comparator)
  Interventions: Other: Manual contact

INTERVENTIONS:
Other: Neck passive mobilizations — Passive mobilizations performed to the neck of the participant by a Physiotherapist
  Arms: Neck passive mobilizations
Other: Manual contact — Manual contact applied to the neck of the participant by a Physiotherapist
  Arms: Manual contact

SUMMARY:
This study investigates the effects of spinal mobilizations on neck symptoms and sympathetic nervous system activity in people with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of neck pain
* Non-traumatic history of onset
* Pain has a clear mechanical aggravating and easing positions or movements
* Limited range of motion
* Local provocation tests produce recognisable symptoms
* A positive expectation that mobilisations will help

Exclusion Criteria:

* No neurological deficit
* No signs of central hyperexcitability
* Referral to other health professional to exclude red flags not required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Global rating of change scale | Immediately after the intervention
  Measures overall improvement as perceived by the participant. It is a 15-point scale ranging from -7 (a very great deal worse), through 0 (no change), to +7 (a great deal better). Values above 0 denote improvement following treatment, 0 denotes no change, and values below 0 denote worsening after the treatment. The higher the value, the greater the improvement; the lower the value, the greater the worsening. The participant will be asked to provide a value that represents their change (they may give 0, which denotes no change) following the intervention.
Change in pain reported by the participant during neck movements | Baseline and immediately after the intervention
  The participant will be asked to report if he/she has pain on each of the following movements: flexion, extension, side flexion and rotation
Change in Sympathetic nervous system activity using skin conductance | Baseline, during the intervention and immediately after the intervention
  Skin conductance in the index and ring finger will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Basque Country, Faculty of Medicine and Infirmary, Leioa, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Undecided